CLINICAL TRIAL: NCT06557941
Title: The Risk Factors of Extubation Failure in Pediatric Intensive Unite Patients at Sohag University Hospitals
Brief Title: Risk Factors of Extubation Failure in PICU Patients
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mariam Rafaat Helmy, postgraduate pediatriacian, Sohag University
Other Study IDs: Soh-Med-24-07-11MS
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Extubation Failure
Keywords: extubation failure; mechanical ventilation; PICU

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: None Retained — Patients will be divided into 2 groups :
  group A : successful extubation. group B : failed extubation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A:successful extubation: mechanically ventilated PICU patients who pass spontaneous breathing trial and air leak test , extubated and not requiring to be re-intubated within 48 hours.
- B: failed extubation: mechanically ventilated PICU patients who don't pass spontaneous breathing trial and air leak test , extubated and requiring to be re-intubated within 48 hours.

SUMMARY:
Up to 20% of MV patients experience EF [10]. EF is defined as the need to reinsert the endotracheal tube to resume MV in patients extubated for less than 48 hours. It has high rates of morbidity and mortality, prolongs the duration of MV and thus causes a longer stay in the PICU and risk of complications such as the need for tracheostomy, the incidence of pneumonia and pulmonary damage, and finally, costs increase as well and death [10, 11] .

DETAILED DESCRIPTION:
Mechanical ventilation (MV) is a common life support modality in 40% of pediatric intensive care unit (PICU) patients. The process of ventilatory support follows a continuum of care, beginning with the patient requiring initial support and ending with the ability to sustain spontaneous breathing [1].

Although MV is a cornerstone in critical care medicine, risks and complications associated with prolonged MV include ventilator associated pneumonia (VAP), barotrauma / volutrauma, decreased cardiac filling, ventilator associated diaphragmatic dysfunction and sepsis [6, 8].

Previous studies recommend extubating patient as early as possible according to clinical course and reversal of the leading causes of intubation. The process of extubation consists of the removal of the endotracheal tube when the patient's physiological status recovers allowing the patient to maintain spontaneous breathing [3,4].

Weaning from MV and extubation are vital steps in patients' recovery; however, these steps are associated with significant risks. Balancing the hazards of premature extubation such as extubation failure (EF) and emergent reintubation with those of prolonged MV is a challenge. [4,5] There is currently a paucity of published evidence-based protocols or guidelines to guide this process; therefore, predictors for successful extubation in critically ill children are not always clear cut. This has resulted in wide variation in practice amongst (PICU) providers that is typically based on institutional norms [4,5, 6]. The most common approach to weaning infants and children is gradual reduction of ventilatory settings not requiring changing the ventilator mode [12].

Up to 20% of MV patients experience EF [10]. EF is defined as the need to reinsert the endotracheal tube to resume MV in patients extubated for less than 48 hours. It has high rates of morbidity and mortality, prolongs the duration of MV and thus causes a longer stay in the PICU and risk of complications such as the need for tracheostomy, the incidence of pneumonia and pulmonary damage, and finally, costs increase as well and death [10, 11] .

At present , several pediatric studies have shown the predictive factors associated with EF ; longer duration of MV ≥7 days and PICU admission ≥ one month , age under one year , malnutrition, respiratory and chronic neurological deterioration , use of sedatives by infusion ≥ 5 days and inotropes ≥ 10 days[6,8] , improper evaluation for extubation readiness , post extubation upper airway obstruction and stridor, residual muscle weakness , pulmonary edema , weak cough reflex[9, 10] , use of uncuffed endotracheal tube , presence of any metabolic and electrolyte imbalances and high ventilator settings prior to extubation [11].

Therapeutic respiratory support, including noninvasive positive pressure ventilation and high-flow nasal cannula, appears to help reduce the need for reintubation in the majority of patients experiencing post extubation respiratory failure. however, Neurologic patients seem to be at higher risk of reintubation despite NIV use [6,13].

Previous researches were carried out in some Egyptian PICUs to investigate the incidence and potential risk factors of EF [1,2,3]. Mahmoud demonstrated that about third of mechanically-ventilated patients in the study experienced EF [2]. Another study showed that the need for longer periods of sedation and high setting on MV in addition to excess tracheal secretions were among strong predictors for EF [3]. Moreover, previous research in our PICU indicated that mortality was high up to 40% [16]. Therefore, investigating the causes of EF in our unit might help in reducing mortality. Furthermore, establishing local protocol of gradual and correct weaning can decrease the risk of EF in our unit.

ELIGIBILITY:
Inclusion Criteria:

* All patient at PICU < 18 years subjected to MV through an endotracheal tube at least >12 hours.
* Patients eligible for weaning from MV according to the weaning criteria (Evidence for some reversal of the underlying cause following for respiratory failure, Adequate oxygenation" PaO2/FIO2 ratio ≥ 200, FIO2 ≤ 0.40, PaO2 ≥ 60, PaCO2 ≤ 60 and PEEP ≤ 5 cmH2O.", PH ≥ 7.25, Respiratory rate (RR) ≤ 45 bpm, Heart rate (HR) ≤ 140 bpm,(rapid shallow breathing index = tidal volume / RR) RSBI ≤ 8 breaths/min/ml/kg body weight, Hemodynamic stable, no or minimal vasopressor or inotropes"[1,12],.
* Appropriate level of consciousness, No continuous sedation infusion nor neuromuscular blocking agents, afebrile, adequate hemoglobin ≥ 7.5 g/dl and/or no evidence of hemorrhage.

Exclusion Criteria:

* Patients less than 30 days.
* Tracheostomized patients.
* Death on mv ≤ 12 hours.
* Unplanned extubation.

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients in PICUS in Sohag University Hospitals.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
successful extubation and weaning from mechanical ventilation | 48 hours
  passing spontaneous trial and air leak test and not requiring to be re-intubated within 2 days
failed extubation , failed weaning from mechanical ventilation | 48 hours
  not passing spontaneous trial and air leak test and not requiring to be re-intubated within 2 days

SECONDARY OUTCOMES:
survival or death | 30 days
  weaning from mechanical ventilation and improvement of the cause of intubation

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Ashry Mohamed, assistant professeer, Study Director — pediatrics department faculty of medicine sohag university; Rania Gamal Mostafa Abdelatif, lecturer, Study Director — pediatrics department faculty of medicine sohag university
Locations (1):
- Sohag University Hospitals, Sohag, Egypt